CLINICAL TRIAL: NCT03762473
Title: Conversion From Tacrolimus to Envarsus in Rapid Metabolizers Post Kidney Transplant Protects Against BK Infection
Brief Title: Conversion to Envarsus Post Kidney Transplant Protects Against BK Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Graham C. Towns, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001068
Record Dates: First submitted 2018-08-27; First posted 2018-12-03 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Renal Transplant Infection
Keywords: Envarsus
MeSH Terms: interventions — Control Groups; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Post transplant patients (kidney transplant alone) with standard of care immunosuppression, no prior rejection, prior BK or opportunistic infection, and negative BK screening at month 1, whom have a concentration/dose of < 1 and a steady state therapeutic level will be eligible. Patients will be converted to envarsus at 20% reduction in dose.
  Interventions: Drug: Study Group
- Control Group (Active Comparator): Post transplant patients (kidney transplant alone) performed between 10-2016 and time of enrollment with standard of care immunosuppression, no prior rejection, prior BK or opportunistic infection, whom had a negative BK screening at month 1 and concentration/dose of < 1 at month 1, and BK data available and month 2,3, 6,9,12.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Study Group — Patients will convert from current tacrolimus dose to an Envarsus dose that is 80% of the total tacrolimus dose. They will take envarsus once daily in the morning and have 24 hour trough levels monitored at the standard of care interval for tacrolimus. Dosing will be titrated to achieve goal levels.
  Other Names: tacrolimus extended-release tablets
  Arms: Study Group
Drug: Control Group — Post transplant patients (kidney transplant alone) performed between 10-2016 and time of enrollment with standard of care immunosuppression, no prior rejection, prior BK or opportunistic infection, whom had a negative BK screening at month 1 and concentration/dose of < 1 at month 1, and BK data available and month 2,3, 6,9,12.
  Other Names: Tacrolimus
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess if the use of Envarsus in place of Tacrolimus-immediate release (IR) in rapid metabolizers post kidney transplant will reduce incidence of BK infection. Efficacy evaluations will include measurement of urine and serum BK values at specified time points and review of any biopsy for BK virus nephropathy. Incidence of rejection, graft failure, and graft dysfunction will also be measured at specified time points.

DETAILED DESCRIPTION:
This will be a single center prospective case control study. The investigators expect 40% of patients will develop BK viruria, 20% BK viremia, 5% BK viral nephropathy (BKVN). Patients will be managed using standard of care for the investigator's center (thymoglobulin induction, tacrolimus/mycophenolate/prednisone). Target tacrolimus level is 8-12 ng/mL for the first 6 months post transplant and 6-9 ng/mL thereafter. BK urine/serum is monitored at 1, 3, 6, 9, 2 months post transplant. A population of 100 patients is calculated to show significant difference for p value < 0.05.

Population:

Study Group: Post transplant patients (kidney transplant alone) with standard of care immunosuppression, no prior rejection, prior BK or opportunistic infection, and negative BK screening at post-transplant month 1, who have a tacrolimus concentration/dose of < 1 and a steady state therapeutic level will be eligible. Patients who consent will be converted to Envarsus at 20% reduction in tacrolimus dose.

Control Group: Post transplant patients (kidney transplant alone performed between 10-2016 and time of enrollment) with standard of care immunosuppression, no prior rejection, prior BK or opportunistic infection, whom had a negative BK screening at post-transplant month 1 and tacrolimus concentration/dose of < 1 at post-transplant month 1, and BK data available for months 2, 3, 6, 9,12 post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age at the time of study entry
* Recipient of a deceased or living donor kidney transplantation
* Maintenance immunosuppression consisting of tacrolimus/ mycophenolate mofetil (MMF)/mycophenolic acid (MPA) (≥1000 mg/720 mg daily) ± prednisone (≤10 mg/day)
* Patient is less than or at 8 weeks post transplant with a negative serum BK Virus screen at 3-4 weeks post transplant
* Patient has a tacrolimus drug dose/concentration of > 1 with therapeutic tacrolimus levels.
* Women of childbearing potential defined as all women physiologically capable of becoming pregnant, must have reviewed Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) and have a negative pregnancy test upon study entry.
* Female (and male) subjects with reproductive potential must agree to use a highly effective method of birth control for the duration of the study. Please note that according to the US product information for MMF/MPA, two reliable forms of contraception must be used simultaneously unless female sterilization, male sterilization, post-menopausal status or total abstinence is the chosen method.

Exclusion Criteria:

* Inability or unwillingness of a patient to give written informed consent or comply with study protocol
* History of graft loss from acute rejection within 1 year after any previous kidney transplant
* History of previous liver, heart, pancreas, or lung transplant
* History of cellular rejection of current allograft prior to enrollment.
* Serum BK virus ≥500 copies/ml by polymerase chain reaction (PCR) at the time of study entry
* Female subjects who are pregnant or breast feeding
* Participation in any other studies with investigational drugs or regimens in the preceding year from the time of study entry
* Any condition or prior treatment which, in the opinion of the investigator, precludes study participation
* Patients requiring the use of azathioprine or a class of drugs that inhibit the mammalian target of rapamycin (mTOR inhibitors)
* Patients with active peptic ulcer disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham C Towns, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 44 | 45
Completed | 43 | 45
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Categorical [Count of Participants; unit: Participants] — Population: the patient who died was not included in the statistics
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 40 | 45 | 85
    >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 50.19 [26 to 68] | 50.19 [26 to 68] | 50.19 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 31 | 30 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 38 | 78
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viruria Results.
Description: The evidence of BK virus infection will be measured by viruria >500 copies.
Time Frame: From baseline to 30 days
Population: data not gathered for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viremia Results.
Description: The evidence of BK virus infection will be measured by viremia >500 copies.
Time Frame: From baseline to 30 days
Population: data not gathered for this time period
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Nephropathy Results.
Description: The evidence of BK virus infection will be measured by nephropathy as defined by Banff classification (sv 40 positivity with or without tubulitis or if/ta).
Time Frame: From baseline to 30 days
Population: data was not gathered at this time period
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viruria Results.
Description: The evidence of BK virus infection will be measured by viruria >500 copies.
Time Frame: From baseline to 120 days
Population: no data was collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viremia Results.
Description: The evidence of BK virus infection will be measured by viremia >500 copies.
Time Frame: From baseline to 120 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Nephropathy Results.
Description: as for outcome 3
Time Frame: From baseline to 120 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viruria Results.
Description: The evidence of BK virus infection will be measured by viruria >500 copies.
Time Frame: From baseline to 210 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viremia Results.
Description: The evidence of BK virus infection will be measured by viremia >500 copies.
Time Frame: From baseline to 210 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Nephropathy Results.
Description: as for outcome 3
Time Frame: From baseline to 210 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Number of Participants With Viruria >500 Copies
Description: Participants will experience less BK infection episodes based on viruria reported with >500 copies.
Time Frame: at 300 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 43 | 45
Participants | 14 | 22

11. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Viremia Results.
Description: The evidence of BK virus infection will be measured by viremia >500 copies.
Time Frame: at 300 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 43 | 45
Participants | 8 | 15

12. Primary Outcome: Participants Will Experience Less BK Infection Episodes Based on Nephropathy Results.
Description: as for outcome 3
Time Frame: at 300 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 43 | 45
Participants | 1 | 1

13. Primary Outcome: Evaluate the Safety of Envarsus Treatment as Assessed by CTCAE v4.0.
Description: Safety will be assessed for all Grade 3 or higher infection
Time Frame: From baseline to 30 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Evaluate the Safety of Envarsus Treatment as Assessed by CTCAE v4.0.
Description: Safety will be assessed for all Grade 3 or higher infection
Time Frame: From baseline to 120 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Evaluate the Safety of Envarsus Treatment as Assessed by CTCAE v4.0.
Description: Safety will be assessed for all Grade 3 or higher infection
Time Frame: From baseline to 210 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Evaluate the Safety of Envarsus Treatment as Assessed by CTCAE v4.0.
Description: Safety will be assessed for all Grade 3 or higher infection
Time Frame: at 300 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 43 | 45
Participants | 1 | 0

17. Secondary Outcome: Evaluate the Effect of Envarsus Conversion as Evidenced by a 15% Decrease in Estimated Glomerular Filtration Rate (GFR) and Proteinuria.
Description: This assessment will include incidence of rejection, graft failure, graft dysfunction as defined by a 15% decrease in estimated glomerular filtration rate (GFR) and proteinuria
Time Frame: From baseline to 30 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Evaluate the Effect of Envarsus Conversion as Evidenced by a 15% Decrease in Estimated Glomerular Filtration Rate (GFR) and Proteinuria.
Description: This assessment will include incidence of rejection, graft failure, graft dysfunction as defined by a 15% decrease in estimated GFR and proteinuria
Time Frame: From baseline to 120 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Evaluate the Effect of Envarsus Conversion as Evidenced by a 15% Decrease in Estimated Glomerular Filtration Rate (GFR) and Proteinuria.
Description: as for outcome 18
Time Frame: From baseline to 210 days
Population: data was not collected for this time period.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Evaluate the Effect of Envarsus Conversion as Evidenced by a 15% Decrease in Estimated Glomerular Filtration Rate (GFR) and Proteinuria.
Description: as for outcome 18
Time Frame: at 300 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 43 | 45
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: at 300 days
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 0/43 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03762473/Prot_SAP_000.pdf